CLINICAL TRIAL: NCT06015984
Title: The Effect of Web-Based Renal Transplantation Nurse Training on Patient-Centered Care Competence and Counseling Skills
Brief Title: Renal Transplantation Nurse Training on Patient-Centered Care Competence and Counseling Skills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Gedik University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EBK-01
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Kidney Transplantation; Nursing; Education; Care; Counseling

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based 8-week Asynchronous Renal Transplantation Nurse Training (Experimental): 1. Week: application of pre-tests
  1. Month: administration of post-tests 3. Month: administration of post-tests
  Interventions: Behavioral: Traning
- non-trained nurse group (No Intervention): 1. Week: application of pre-tests
  1. Month: administration of post-tests 3. Month: administration of post-tests

INTERVENTIONS:
Behavioral: Traning — In order to participate in the training module, a user name and password will be given to the initiative group, the link to be used in the self-managed and asynchronous training platform will be shared, and it will be ensured that it participates in the web-based nurse training, and the training will last for eight weeks.
  Arms: Web-Based 8-week Asynchronous Renal Transplantation Nurse Training

SUMMARY:
There are two main treatments for end-stage renal disease (ESRD): dialysis and transplantation.Renal transplantation is the best and most preferred treatment for ESRD patients.Self management after renal transplantation is difficult. Individuals need appropriate care,education, counseling and support in order to change their behavior to cope with health problems during the transplantation process.The aim of nursing care and education is to enable the individual to acquire the knowledge, skills and attitude to independently carry out daily life activities and to adopt this as a lifestyle.Nursing care and education requires an interdisciplinary teamwork, and in this process, the nurse plays a key role as she constantly interacts with the donor, recipient and family.The research was designed as a randomized controlled experimental study with pretest-posttest design.A total of 60 nurses, 30 in the control group and 30 in the intervention group,who met the criteria for inclusion in the study, will form the sample of the study.After obtaining consent from the nurses in the intervention and control groups, they will be asked to fill out the Nurse InformationForm, the Patient-Centered Care Competency Scale and the Nurses Counseling Skills Scale. Aftercompleting the web-based training, intervention group nurses will be asked to fill in the Patient Centered Care Competency Scale and the Counseling Skills in Nurses Scale at the 1st and 3rd months. No training will be given to the nurses in the control group and they will be asked to fill the Patient-Centered Care Competency Scale and the Counseling Skills for Nurses Scale again.

DETAILED DESCRIPTION:
There are two main treatments for end-stage renal disease (ESRD): dialysis and transplantation. Renal transplantation (RTx) is the best and most preferred treatment for ESRD patients. A successful RTx, made from a living or cadaver donor, improves the quality of life compared to dialysis and fully fulfills the function of the kidney.Self-management after renal transplantation is difficult. Individuals need appropriate care, education, counseling and support in order to change their behavior to cope with health problems during the transplantation process. The aim of nursing care and education is to enable the individual to acquire the knowledge, skills and attitude to independently carry out daily life activities and to adopt this as a lifestyle. Nursing care and education requires an interdisciplinary teamwork, and in this process, the nurse plays a key role as she constantly interacts with the donor, recipient and family.Today, technology-based methods are used to increase compliance with transplantation and are increasingly seen as valuable tools. The aim of this research is to develop and implement a web-based nurse training program for renal transplantation nurses and to examine the effect of this training on nurses' patient-centered care competence and counseling skills. The research was designed as a randomized controlled experimental study with pretest-posttest design.

The population of the research will be 1870 nurses registered to the Turkish Nephrology, Dialysis and Transplantation Nurses Association. A total of 60 nurses, 30 in the control group and 30 in the intervention group, who met the criteria for inclusion in the study, will form the sample of the study.The research will be carried out on the website www.bobreknakliokulu.com, which will be developed after a preliminary interview with the nurses working in the renal transplantation clinics between April and August 2023, and they will be included in the web-based training as self-managed and asynchronous for 8 weeks.After obtaining consent from the nurses in the intervention and control groups, they will be asked to fill out the Nurse Information Form, the Patient-Centered Care Competency Scale and the Nurses Counseling Skills Scale. After completing the web-based training, intervention group nurses will be asked to fill in the Patient-Centered Care Competency Scale and the Counseling Skills in Nurses Scale at the 1st and 3rd months. No training will be given to the nurses in the control group and they will be asked to fill the Patient-Centered Care Competency Scale and the Counseling Skills for Nurses Scale again.It is expected that the renal transplantation nurses who receive this training will contribute positively to the increase of evidence-based knowledge and the development of clinical practices, the competence of patient-centered care and the management of counseling skills in line with clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Having a maximum of 3 years of working experience in the Renal Transplantation clinic
* Having a bachelor's degree in nursing

Exclusion Criteria:

* Nurses not completing all web-based nursing education modules
* It will be caused by nurses not completing the 20-minute website usage period determined for each training module.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient-Centered Care Competency Scale | 3 months
  Scale, by Hwang (2015); It was developed in order to determine the competencies of nurses in patient-centered care. The Turkish validity and reliability of the scale was made by Arslanoğlu and Kırılmaz (2019). The Cronbach Alpha coefficient is 0.850. Patient-centered care competence consists of 17 questions and 4 sub-dimensions. Sub-dimensions; respecting the point of view (perspective) of patients (item 1-6), encouraging patient participation in care processes (items 7 and 11), ensuring patient comfort (items 12 and 14), and defending the rights of patients (15. - Article 17). Scale; It was designed as a 5-point Likert scale: 1-Strongly Disagree, 2-Disagree, 3-Undecided, 4-Agree, 5-Strongly Agree.

SECONDARY OUTCOMES:
Counseling Skills Scale for Nurses | 3 months
  After the item pool created by Avcı and Kumcagiz in 2019 was finalized, it was applied to 204 nurses for explanatory factor analysis. The scale consists of 10 items and is a single factor. Afterwards, confirmatory factor analysis (CFA) was performed on 200 nurses. With confirmatory factor analysis, the fit index values of the single factor structure were found to be within acceptable limits (χ2=94,785, sd=33, χ2/sd= 2.872, RMSEA=0.097, GFI=0.92, AGFI=0.86, CFI=0.92 and IFI=0.92) . The validity of the scale was examined by performing EFA and CFA. The reliability of the scale was examined with Cronbach's alpha coefficient and Split-half. Cronbach alpha was calculated as 0.88 and Split-half as 0.86.

CONTACTS AND LOCATIONS:
Overall Officials: Emek Bakanoğlu Kalkavan, Principal Investigator — Istanbul Gedik University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiaranai C. The Lived Experience of Patients Receiving Hemodialysis Treatment for End-Stage Renal Disease: A Qualitative Study. J Nurs Res. 2016 Jun;24(2):101-8. doi: 10.1097/jnr.0000000000000100. PMID 26275156
- [Background] Samarehfekri A, Dehghan M, Arab M, Ebadzadeh MR. Effect of Foot Reflexology on Pain, Fatigue, and Quality of Sleep after Kidney Transplantation Surgery: A Parallel Randomized Controlled Trial. Evid Based Complement Alternat Med. 2020 Aug 1;2020:5095071. doi: 10.1155/2020/5095071. eCollection 2020. PMID 32831868
- [Background] Mathes T, Grosspietsch K, Neugebauer EAM, Pieper D. Interventions to increase adherence in patients taking immunosuppressive drugs after kidney transplantation: a systematic review of controlled trials. Syst Rev. 2017 Nov 29;6(1):236. doi: 10.1186/s13643-017-0633-1. PMID 29187249
- [Background] Kleber J, Cohen B. Reducing Waste and Increasing Sustainability in Health Care Settings. Am J Nurs. 2020 Apr;120(4):45-48. doi: 10.1097/01.NAJ.0000660032.02514.ec. PMID 32218047
- [Background] Kohler B, Kellerer C, Schultz K, Wittmann M, Atmann O, Linde K, Hapfelmeier A, Schneider A. An Internet-Based Asthma Self-Management Program Increases Knowledge About Asthma. Dtsch Arztebl Int. 2020;117(5):64-71. doi: 10.3238/arztebl.2020.0064. PMID 32070472
- [Background] Coresh J, Hu JR, Bello AK, Feldman HI, Fogo AB, Ganji MR, Harris DC, Levey AS, Okpechi IG, Stengel B, Thomas B, Wiecek A, Gansevoort RT. Action plan for determining and monitoring the prevalence of chronic kidney disease. Kidney Int Suppl (2011). 2017 Oct;7(2):63-70. doi: 10.1016/j.kisu.2017.07.002. Epub 2017 Sep 20. PMID 30675421
- [Background] Chisholm-Burns M, Pinsky B, Parker G, Johnson P, Arcona S, Buzinec P, Chakravarti P, Good M, Cooper M. Factors related to immunosuppressant medication adherence in renal transplant recipients. Clin Transplant. 2012 Sep-Oct;26(5):706-13. doi: 10.1111/j.1399-0012.2011.01589.x. Epub 2012 Feb 10. PMID 22324912
- [Background] Zala P, Schmid-Mohler G. Patients' Experiences of a Nurse-Led Self-Management Intervention After Kidney Transplantation. Nephrol Nurs J. 2022 Jan-Feb;49(1):45-57. PMID 35225495
- [Background] Horka K. Optimizing Care in Kidney Transplantation. Crit Care Nurs Clin North Am. 2022 Dec;34(4):443-451. doi: 10.1016/j.cnc.2022.08.003. Epub 2022 Oct 12. PMID 36336434